CLINICAL TRIAL: NCT05701891
Title: The (Cost-)Effectiveness of an Innovative, Personalised Intervention of Therapeutic VirtuAl Reality IntEgrated Within physioTherapY for a Subgroup of Complex Chronic Low Back Pain Patients
Brief Title: Virtual Reality Integrated Within Physiotherapy for Patients With Complex Chronic Low Back Pain
Acronym: VARIETY
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: HAN University of Applied Sciences (Other)
Responsible Party: Principal Investigator, Bart Staal, Professor (lector), HAN University of Applied Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 10270032021502
Record Dates: First submitted 2022-12-02; First posted 2023-01-27 (Actual); Last update posted 2023-04-14 (Actual); Status verified 2023-04

CONDITIONS: Chronic Low-back Pain
Keywords: Chronic low back pain; Chronic pain
MeSH Terms: conditions — Chronic Pain | interventions — Physical Therapy Modalities

STUDY DESIGN:
Intervention Model Description: This study is a two-arm cluster-randomized controlled trial. Twenty physiotherapists with expertise in chronic LBP treatment will be recruited and equally randomised (10 in each arm) on the level of physiotherapy practice using allocation concealment. This clustered design means that eligible patients consulting a participating physiotherapist will be automatically allocated to the study arm (experimental or control arm) to which the physiotherapy practice was allocated.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Physiotherapy with integrated VR (Experimental): Our intervention will be a 12-week personalised, VR-integrated physiotherapy intervention in which a selection of existing VR modules developed by our partners (i.e. Reducept and SyncVR) will be integrated into physiotherapy treatment. The following VR modules will be used: education (Reducept), relaxation and distraction (SyncVR Relax & Distract), activation (SyncVR Fit). Patients will use the Pico Neo 3 VR headset at the physiotherapy practice and at home 5 days a week for 10-30 minutes. In addition, physiotherapists will help patients transition from movements performed in a VR context to daily activities without VR.
  Interventions: Combination Product: Physiotherapy with integrated Virtual Reality
- Physiotherapy (usual care) (Active Comparator): The control condition is usual physiotherapy care for 12 weeks.
  Interventions: Other: Physiotherapy (usual care)

INTERVENTIONS:
Combination Product: Physiotherapy with integrated Virtual Reality — A 12-week personalised, VR-integrated physiotherapy intervention.
  Other Names: Reducept; SyncVR Relax & Distract; SyncVR Fit
  Arms: Physiotherapy with integrated VR
Other: Physiotherapy (usual care) — A 12-week usual physiotherapy care intervention.
  Arms: Physiotherapy (usual care)

SUMMARY:
This study examines the effect of a 12-week intervention of physiotherapy with integrated Virtual Reality (VR) on 120 patients with complex chronic low back pain. Patients in the intervention group will receive physiotherapy with integrated VR, while patients in the control group will receive physiotherapy as usual. The (cost-)effectiveness of this intervention will be investigated at 3 months and 12 months follow-up.

DETAILED DESCRIPTION:
Rationale: Physiotherapy, mainly consisting of exercise therapy and patient education, is a first-choice primary care treatment for patients with chronic low back pain (LBP), but unfortunately, especially patients with severe disability and pain demonstrate poor outcomes. Therapeutic VR is considered a potential breakthrough for LBP patients in general and for our complex group of patients with severe disability and pain in particular, as it specifically targets the identified limitations of usual physiotherapy. Therefore, a personalised, VR-integrated physiotherapy intervention, tailored to specific patient characteristics, is expected to result in larger improvements in physical functioning and pain, and more favourable cost-effectiveness, compared to usual physiotherapy.

Objective: The primary objective is to investigate whether a personalised, physiotherapy intervention with integrated therapeutic virtual reality (VR) is (cost-)effective at 3 months and 12 months follow-up, compared to usual physiotherapy, in a subgroup of patients with complex chronic low back pain (LBP) and severe disability and pain.

Study design: Cluster randomised controlled trial.

Study population: 120 chronic LBP patients with combination of severe disability and severe pain, consulting a physiotherapist in primary care.

Intervention: The experimental intervention will be a 12-week personalised, VR-integrated physiotherapy intervention in which a selection of existing VR modules developed by research partners (i.e. Reducept and SyncVR) will be integrated into physiotherapy based on the recommendations of the LBP guidelines. The control intervention will be physiotherapy as usual.

Main study parameters/endpoints: Physical functioning (primary outcome), in addition to pain and a minimal set of other secondary clinical, adherence-related, psychological and economic measures, at baseline and 1, 3 and 12 months follow-up.

ELIGIBILITY:
Inclusion Criteria:

* LBP > 3 months as reason to visit physiotherapist
* absence of 'red flags' or signs of specific LBP
* combination of severe disability (Oswestry Disability Index (ODI) score ≥ 30) and severe pain (numeric rating score (NRS) ≥ 5)
* age 18-80 years
* provides informed consent.

Exclusion Criteria:

* severe (physical or mental) comorbidity that will substantially hinder the physiotherapy
* planned diagnostic or invasive therapeutic procedure (e.g. injection, nerve block or operation) for LBP in next three months
* no comprehension of Dutch language
* inability to use VR (e.g. epilepsy, open wounds on face or severe visual impairment)
* no email-address and Wi-Fi

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2024-03 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Change in physical functioning measured using the Oswestry Disability Index (ODI) | baseline, 1, 3 and 12 months
  This questionnaire on physical functioning scores from 0 (best possible score) to 100 (worst possible score).

SECONDARY OUTCOMES:
Change in pain intensity measured using the Numeric Pain Rating Scale (NPRS) | baseline, 1, 3 and 12 months
  This questionnaire on pain intensity scores from 0 (best possible score) to 10 (worst possible score).
Change in pain-related fears measured using the Fear-Avoidance Beliefs Questionnaire - Physical Activity (FABQ-PA) | baseline, 1, 3 and 12 months
  The FABQ scores from 0 (best possible score) to 30 (worst possible score).
Change in pain-related fears measured using the Pain Catastrophizing Scale (PCS) | baseline, 1, 3 and 12 months
  The PCS scores from 0 (best possible score) to 52 (worst possible score).
Change in physical activity on self-reported moderate physical activity (i.e. minutes of performed physical activity in past week) | baseline, 1, 3 and 12 months
  This questionnaire scores from 0 minutes (worst possible score) to 1680 minutes (best possible score, based on a maximum of 4 hours of possible moderate physical activity per day).
Change in general effect measured using the Global Perceived Effect (GPE) | baseline, 1, 3 and 12 months
  This questionnaire scores from 0 (worst possible score) to 14 (best possible score).
Change in problems with activities measured using the Patient Specific Complaints (PSK) | baseline and 3 months
  This questionnaire scores from 0 (best possible score) to 10 (worst possible score) per activity.
Change in pain self-efficacy measured using the Pain Self-Efficacy Questionnaire (PSEQ) | baseline, 1, 3 and 12 months
  This questionnaire scores from 0 (worst possible score) to 60 (best possible score).
Change in cost-effectiveness measured using the EuroQol - 5 Dimensions - 5 Level (EQ-5D-5L) | baseline, 1, 3, 6 and 12 months
  The questionnaire consists of two components: the EQ-5D descriptive system and the EQ Visual Analogue Scale (EQ-VAS).The first part consists of five subjects, from which for each subject a single EQ-5D index score can be calculated ranging from 0 (worst possible score) to 1 (best possible score). The EQ-VAS scores from 0 (worst possible score) to 100 (best possible score).

CONTACTS AND LOCATIONS:
Locations (1):
- HAN University of Applied Sciences, Nijmegen, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Slatman S, Ostelo R, van Goor H, Staal JB, Knoop J. Physiotherapy with integrated virtual reality for patients with complex chronic low back pain: protocol for a pragmatic cluster randomized controlled trial (VARIETY study). BMC Musculoskelet Disord. 2023 Feb 20;24(1):132. doi: 10.1186/s12891-023-06232-0. PMID 36803315

DOCUMENTS (1):
  • Statistical Analysis Plan (2023-01-27): https://cdn.clinicaltrials.gov/large-docs/91/NCT05701891/SAP_000.pdf